CLINICAL TRIAL: NCT01399593
Title: A Randomized, Open-label, Multicenter Trial to Determine Safety and Efficacy of Eculizumab in the Prevention of Antibody Mediated Rejection (AMR) in Living Donor Kidney Transplant Recipients Requiring Desensitization Therapy
Brief Title: Safety & Efficacy of Eculizumab to Prevent AMR in Living Donor Kidney Transplant Recipients Requiring Desensitization
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not achieve statistical significance for primary endpoint
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C10-001; 2010-019630-28 (EudraCT Number); BB-IND: 100,003 (Other: FDA IND: 100,003)
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Antibody Mediated Rejection
Keywords: Antibody Mediated Rejection; AMR; Acute Humoral Rejection; AHR; Living Donor; Kidney Transplant
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eculizumab (Experimental): Patients were to receive eculizumab 1200 mg prior to allograft transplantation (Day 0, starting approximately one hour prior to kidney allograft reperfusion), eculizumab 900 mg (Days 1, 7, 14, 21, and 28), and eculizumab 1200 mg (Weeks 5, 7 and 9). All doses of eculizumab were administered intravenously: the median infusion time was 39 minutes.
  Interventions: Drug: Eculizumab
- Standard of Care (No Intervention): Patients received standard of care (SOC) prophylactic therapy for acute AMR according to the SOC choice at each participating investigative site, which could have included any combination of plasmapheresis (PP) and intravenous immunoglobulin (IVIg). Patients randomized to SOC who were diagnosed with AMR could have received eculizumab for the treatment of AMR after initially receiving PP and/or IVIg.

INTERVENTIONS:
Drug: Eculizumab
  Other Names: Soliris
  Arms: Eculizumab

SUMMARY:
The purpose of this trial was to determine the safety and efficacy of eculizumab in the prevention of antibody-mediated rejection (AMR) in sensitized recipients of a living donor kidney transplant requiring desensitization therapy.

DETAILED DESCRIPTION:
The main objective of this study was to evaluate the safety and efficacy of eculizumab to prevent AMR in sensitized recipients of living donor kidney transplants requiring desensitization therapy prior to transplantation. The primary endpoint focused on acute AMR during the first 9 weeks post-transplantation.

Patients were to be vaccinated against N. meningitidis at least 14 days prior to study drug initiation and revaccinated 30 days later. If not vaccinated 14 days prior, prophylactic antibiotics were to be administered. Pre-transplant infectious disease assessment was to be performed as part of the screening assessment.

Patients were to undergo desensitization therapy according to the practice of the local transplant center prior to transplantation, and this desensitization practice was to be uniformly applied for all patients at that center throughout the study. The actual length of desensitization for an individual patient was based on the clinical judgment of the Transplant Center team. Rituximab was prohibited in all patients as part of the pre-transplantation desensitization therapy due to potential pharmacodynamic interactions.

The control group was designed to test eculizumab against the best available care (referred to as standard of care, or SOC) consisting of plasmapheresis (PP) and/or intravenous immunoglobulin (IVIg). The best available care consisting of PP and IVIg was chosen because these modalities combined represented the most prevalent therapy reported in the literature and were the best available therapies at the time of this protocol's inception as per the transplant community.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old
2. Patients with Stage IV or Stage V chronic kidney disease who will receive a kidney transplant from a living donor to whom they are sensitized and require desensitization prior to transplantation

Exclusion Criteria:

1. ABO incompatible with living donor
2. Any medical condition that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confounds the assessment of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-11-02 (Actual); Primary Completion 2014-05-13 (Actual); Study Completion 2015-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masayo Ogawa, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (39):
- United States (17):
  - Birmingham, Alabama
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Livingston, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Houston, Texas
- Australia (4):
  - North Terrace, South Australia
  - Camperdown
  - Clayton VIC
  - Parkville VIC
- France (3):
  - Paris
  - Toulouse
  - Tours
- Germany (2):
  - Dresden
  - Heidelberg
- Italy (2):
  - Milan
  - Padua
- Rotterdam, Netherlands
- Oslo, Norway
- Barcelona, Spain
- Sweden (3):
  - Gothenburg
  - Huddinge
  - Uppsala
- United Kingdom (5):
  - London, England
  - Oxford, England
  - Birmingham
  - Cambridge
  - Coventry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marks WH, Mamode N, Montgomery RA, Stegall MD, Ratner LE, Cornell LD, Rowshani AT, Colvin RB, Dain B, Boice JA, Glotz D; C10-001 Study Group. Safety and efficacy of eculizumab in the prevention of antibody-mediated rejection in living-donor kidney transplant recipients requiring desensitization therapy: A randomized trial. Am J Transplant. 2019 Oct;19(10):2876-2888. doi: 10.1111/ajt.15364. Epub 2019 Apr 19. PMID 30887675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period lasted from Nov 2011 to Mar 2014. Forty-one sites in Australia, the European Union, and North America participated in this study.
Pre-assignment Details: Written consent was provided prior to performing any study-required assessments (N = 275). Patients who passed screening (N = 137) underwent desensitization therapy according to local transplant center practice prior to transplantation. A total of 104 patients were randomized; of these, 102 were transplanted and received eculizumab or SOC.
Groups:
- Eculizumab: Patients were to receive eculizumab 1200 mg prior to allograft transplantation (Day 0, starting approximately one hour prior to kidney allograft reperfusion), eculizumab 900 mg (Days 1, 7, 14, 21, and 28), and eculizumab 1200 mg (Weeks 5, 7 and 9).
Period: Overall Study
Arm/Group | Eculizumab | Standard of Care
Started | 51 | 51
Completed | 48 | 49
Not Completed | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 1
Not completed — Transplantectomy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Eculizumab: Patients in the eculizumab treatment group were to receive eculizumab for 9 weeks according to the following dosing regimen:
  Eculizumab 1200 mg prior to allograft transplantation (Day 0, starting approximately one hour prior to kidney allograft reperfusion), eculizumab 900 mg (Days 1, 7, 14, 21, and 28), and eculizumab 1200 mg (Weeks 5, 7 and 9). All doses of eculizumab were administered intravenously.
- Standard of Care (SOC): Patients in the standard of care (SOC) treatment group received prophylactic therapy for acute AMR according to the SOC choice at each participating investigative site, which could have included any combination of plasmapheresis (PP) and intravenous immunoglobulin (IVIg). Patients randomized to SOC who were diagnosed with AMR could have received eculizumab for the treatment of AMR after initially receiving PP and/or IVIg.
- Total: Total of all reporting groups
Arm/Group | Eculizumab | Standard of Care (SOC) | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn - gestational age < 37 wk | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 47 | 49 | 96
  From 65 to 84 years | 4 | 2 | 6
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 30 | 67
  Male | 14 | 21 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patients appearing under "Unknown or Not Reported" were categorized as "Other" by the investigator.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 6 | 12
    White | 37 | 36 | 73
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 1 | 5
  France | 3 | 7 | 10
  Germany | 1 | 1 | 2
  Italy | 2 | 4 | 6
  Netherlands | 0 | 3 | 3
  Norway | 1 | 1 | 2
  Spain | 3 | 4 | 7
  Sweden | 1 | 4 | 5
  United Kingdom | 10 | 5 | 15
  United States | 26 | 21 | 47
Total Donor-Specific Antibodies (DSA) [Mean (Standard Deviation); unit: mean fluorescence intensity (MFI)] — The presence of donor-specific antibodies (DSA) indicates that a patient has become sensitized, i.e., has preformed antibodies against donor specific human leukocyte antigens (HLAs). A higher DSA level indicates greater sensitization and greater risk of antibody-mediated rejection (AMR). Population: Data unavailable for 4 subjects.
  mean fluorescence intensity (MFI)
    number analyzed (Participants) | 50 | 48 | 98
    (all) | 15394.7 (14163.78) | 17469.8 (12573.44) | 16411.1 (13380.16)
Highest Single Donor-Specific Antibodies (DSA) [Mean (Standard Deviation); unit: mean fluorescence intensity (MFI)] — The presence of donor-specific antibodies (DSA) indicates that a patient has become sensitized, i.e., has preformed antibodies against donor specific human leukocyte antigens (HLAs). A higher DSA level indicates greater sensitization and greater risk of antibody-mediated rejection (AMR). Population: Data unavailable for 4 subjects.
  mean fluorescence intensity (MFI)
    number analyzed (Participants) | 50 | 48 | 98
    (all) | 8135 (4048.08) | 8740.7 (4289.97) | 8431.7 (4157.87)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure Rate
Description: The primary efficacy variable was a binary outcome variable where patients meeting the composite endpoint of the occurrence of 1) biopsy-proven acute AMR, 2) graft loss, 3) patient death, or 4) loss to follow-up definition at Week 9 post-transplantation were considered treatment failures and all others were considered treatment successes.
Time Frame: 9 weeks post-transplantation
Population: Full analysis set, defined as patients who were randomized, received a living donor kidney transplant, and were treated (either with eculizumab or SOC), based on randomized treatment groups.
Measure: Count of Participants; unit: Participants
Groups:
- Eculizumab: Patients were to receive eculizumab 1200 mg prior to allograft transplantation (Day 0, starting approximately one hour prior to kidney allograft reperfusion), eculizumab 900 mg (Days 1, 7, 14, 21, and 28), and eculizumab 1200 mg (Weeks 5, 7 and 9). All doses of eculizumab were administered intravenously.
- Standard of Care: Patients in the standard of care (SOC) treatment group received prophylactic therapy for acute AMR according to the SOC choice at each participating investigative site, which could have included any combination of plasmapheresis (PP) and intravenous immunoglobulin (IVIg). Patients randomized to SOC who were diagnosed with AMR could have received eculizumab for the treatment of AMR after initially receiving PP and/or IVIg.
Arm/Group | Eculizumab | Standard of Care
Number analyzed (Participants) | 51 | 51
Participants | 5 | 7
Statistical Analysis 1: Comparison: Eculizumab vs Standard of Care; Test type: Superiority; p = 0.76, Fisher Exact; Proportion difference = -3.9, 95% CI 2-sided [-23.9 to 16.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 3-year study period.
Arm/Group | Eculizumab | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/51 | 1/51
Serious Adverse Events (participants affected / at risk) | 43/51 | 48/51
Other Adverse Events (participants affected / at risk) | 51/51 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=51) | Standard of Care (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac perforation (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Diverticulum (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 0
Hypothermia (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 22 | 28
Abdominal sepsis (Infections and infestations) | 1 | 0 — Fatality occurred in one patient who experienced both one serious adverse event of abdominal sepsis on Day 16 and one serious adverse event of bacterial sepsis on Day 36.
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 — Fatality occurred in one patient who experienced both one serious adverse event of abdominal sepsis on Day 16 and one serious adverse event of bacterial sepsis on Day 36.
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 4 | 6
Gastroenteritis (Infections and infestations) | 0 | 4
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 2
Giardiasis (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 4 | 2
Renal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 7
Urinary tract infection bacterial (Infections and infestations) | 2 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 2
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 4 | 2
Wound infection (Infections and infestations) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Ateriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 1
Delayed graft function (Injury, poisoning and procedural complications) | 2 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Anti-glomerular basement membrane antibody (Investigations) | 1 | 0
Antibody test positive (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1
Drug level increased (Investigations) | 1 | 0 — High level of tacrolimus
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 2 | 3
Nephrectasia (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 1
Ureteric dilatation (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Convalescent (Social circumstances) | 1 | 0
Nephrostomy (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 3 | 5
Superior vena cava occlusion (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=51) | Standard of Care (N=51)
Anaemia (Blood and lymphatic system disorders) | 16 | 28
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 16 | 23
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 12
Tachycardia (Cardiac disorders) | 6 | 10
Vision blurred (Eye disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 13
Abdominal pain lower (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 14 | 15
Diarrhoea (Gastrointestinal disorders) | 22 | 27
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Flatulence (Gastrointestinal disorders) | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 26 | 19
Vomiting (Gastrointestinal disorders) | 13 | 7
Asthenia (General disorders) | 10 | 10
Chest pain (General disorders) | 7 | 3
Chills (General disorders) | 2 | 5
Influenza like illness (General disorders) | 2 | 3
Malaise (General disorders) | 1 | 3
Oedema (General disorders) | 5 | 5
Oedema peripheral (General disorders) | 15 | 21
Pain (General disorders) | 5 | 7
Pyrexia (General disorders) | 12 | 16
Drug hypersensitivity (Immune system disorders) | 5 | 3
Kidney transplant rejection (Immune system disorders) | 19 | 17
BK virus infection (Infections and infestations) | 12 | 9
Bronchitis (Infections and infestations) | 4 | 2
Cellulitis (Infections and infestations) | 2 | 3
Cytomegalovirus infection (Infections and infestations) | 2 | 4
Cytomegalovirus viraemia (Infections and infestations) | 6 | 3
Escherichia urinary tract infection (Infections and infestations) | 4 | 3
Gastroenteritis (Infections and infestations) | 5 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 8
Oral candidiasis (Infections and infestations) | 5 | 2
Pneumonia (Infections and infestations) | 0 | 4
Respiratory tract infection (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 13 | 11
Urinary tract infection (Infections and infestations) | 28 | 18
Urinary tract infection bacterial (Infections and infestations) | 5 | 1
Urinary tract infection enterococcal (Infections and infestations) | 4 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 | 1
Incision site pain (Injury, poisoning and procedural complications) | 8 | 6
Perinephric collection (Injury, poisoning and procedural complications) | 3 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Procedural pain (Injury, poisoning and procedural complications) | 7 | 8
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 6
Wound secretion (Injury, poisoning and procedural complications) | 0 | 4
Antibody test positive (Investigations) | 3 | 0
Blood creatinine increased (Investigations) | 9 | 12
Liver function test abnormal (Investigations) | 7 | 5
Weight decreased (Investigations) | 2 | 3
Weight increased (Investigations) | 5 | 4
Acidosis (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 9
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 2
Fluid overload (Metabolism and nutrition disorders) | 4 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 15
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 14 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 16 | 12
Metabolic acidosis (Metabolism and nutrition disorders) | 12 | 10
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 8
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Nervous system disorders) | 7 | 6
Headache (Nervous system disorders) | 14 | 9
Migraine (Nervous system disorders) | 4 | 2
Tremor (Nervous system disorders) | 14 | 14
Anxiety (Psychiatric disorders) | 8 | 6
Depression (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 7 | 11
Acute kidney injury (Renal and urinary disorders) | 4 | 3
Anuria (Renal and urinary disorders) | 0 | 4
Bladder spasm (Renal and urinary disorders) | 3 | 2
Dysuria (Renal and urinary disorders) | 3 | 4
Haematuria (Renal and urinary disorders) | 5 | 10
Nocturia (Renal and urinary disorders) | 3 | 0
Oliguria (Renal and urinary disorders) | 2 | 6
Polyuria (Renal and urinary disorders) | 6 | 4
Proteinuria (Renal and urinary disorders) | 9 | 6
Renal impairment (Renal and urinary disorders) | 4 | 2
Renal tubular necrosis (Renal and urinary disorders) | 2 | 4
Urinary retention (Renal and urinary disorders) | 1 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 9
Rash (Skin and subcutaneous tissue disorders) | 5 | 3
Deep vein thrombosis (Vascular disorders) | 4 | 1
Haematoma (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 13 | 15
Hypotension (Vascular disorders) | 8 | 11
Lymphocele (Vascular disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
Data interpretation confounded by open-label study with potential reporting bias, unequal exposure to randomized prevention therapy between groups, some patients in SOC arm received eculizumab for treatment of AMR, all patients immunosuppressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No